CLINICAL TRIAL: NCT06526312
Title: Testing Technology-Based Implementation Strategies for a Family-Based Pediatric Health Behavior Intervention in Community-Based Primary Care: A Cluster Randomized Factorial Trial
Brief Title: Primary Care Evidence-based Approach for Improving Lifelong Health
Acronym: PREVAIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Northwestern University (Other); University of Oregon (Other); University of Utah (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R61HL166976 (NIH)
Record Dates: First submitted 2024-07-12; First posted 2024-07-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Clinical Trial
Keywords: implementation; cost-effectiveness; health behaviors; BMI
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: We will test the hypotheses related to implementation strategies at α=.025 to control the family-wise type I error rate at 0.05: (1) mean difference in fidelity in favor of those randomized to the fidelity support condition (including Lyssn, COACH coding, and group supervision), (2) higher engagement for those randomized to SMS. Each hypothesis will be tested under the framework of a linear mixed-effects model to account for care team, FCU4Health Coordinator, and family-level clustering. In addition to the main, each model will include random effects for care team and Coordinator, and covariates used in the restricted randomization. Updated power analyses were performed by simulation assuming 80% complete data for Lyssn and COACH scores (fidelity strategy) and 95% data available on SMS text messaging (i.e., allowing for up to a very conservative 5% opt-out rate).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SMS/Text (CAMPI) (Experimental): Receives interactive content with prompts via SMS (text) message to participant cellular phones developed within this project using the CAMPI platform.
  Interventions: Behavioral: SMS/Text (CAMPI); Behavioral: Family Check-Up 4 Health (FCU4Health)
- Fidelity Monitoring (Lyssn and COACH) (Experimental): Standard Training Activities
  1. asynchronous training in the program via an e-learning program
  2. synchronous training led by a certified FCU4Health Trainer Standard Supervision Activities
  3. use of the valid and reliable COACH observational fidelity rating system to provide individualized feedback from COACH ratings to BHCs
  4. group supervision (typically for a period of a year provided by a certified Trainer and then taken over by the organization in a train-the-trainer type model) Enhanced Supervision Activities
  5. use of the Lyssn system to provide individualized feedback to BHCs
  All BHCs will receive the standard training activities (a-b). For the experimental condition, half of the BHCs will be randomly assigned to full fidelity support strategy, which will include the standard and enhanced supervision activities (c-e).
  Interventions: Behavioral: Fidelity Monitoring (Lyssn and COACH); Behavioral: Family Check-Up 4 Health (FCU4Health)
- SMS/Text (CAMPI) and Fidelity Monitoring System (Lyssn and COACH) (Experimental): Receives interactive content with prompts via SMS (text) message to participant cellular phones developed within this project using the CAMPI platform.
  Receives fidelity monitoring via COACH and Lyssn.
  Interventions: Behavioral: SMS/Text (CAMPI); Behavioral: Fidelity Monitoring (Lyssn and COACH); Behavioral: Family Check-Up 4 Health (FCU4Health)
- No CAMPI or Fidelity Monitoring (Experimental): Receives neither SMS/Text (CAMPI) or Fidelity Monitoring (Lyssn and COACH).
  Interventions: Behavioral: Family Check-Up 4 Health (FCU4Health)

INTERVENTIONS:
Behavioral: SMS/Text (CAMPI) — Configurable Assessment Messaging Platform for Interventions (CAMPI) is a SMS text messaging platform to promote motivation and home practice.
  Arms: SMS/Text (CAMPI); SMS/Text (CAMPI) and Fidelity Monitoring System (Lyssn and COACH)
Behavioral: Fidelity Monitoring (Lyssn and COACH) — Lyssn's HIPAA-compliant, cloud-based platform uses embedded speech-to-text transcription from audio recorded sessions for rapid assessment and easy session review for supervisors and interventionists.
  The COACH fidelity rating system assesses clinical skills in five domains considered essential for the effective provision of the FCU and the EDP intervention sessions. The COACH rating form is used to assess the extent to which the provider is:
  Conceptually accurate and adherent to the intervention model Observant and responsive to the family's needs Active in structuring the session Careful when teaching and providing feedback Helpful in building hope and motivation
  Arms: Fidelity Monitoring (Lyssn and COACH); SMS/Text (CAMPI) and Fidelity Monitoring System (Lyssn and COACH)
Behavioral: Family Check-Up 4 Health (FCU4Health) — An evidence-based, data-driven, individually tailored parenting intervention with evidence of effectiveness on child and family health behaviors and psychosocial well-being. The program includes three components: 1) a comprehensive family assessment, 2) feedback and motivation session, and 3) individually tailored follow-up support (including parent training modules from the Everyday Parenting curriculum and connection with community resources). Dosage and content of these follow-up sessions are driven by the results of the assessment and family interest. The assessment, feedback and motivation session, and follow-up support are repeated annually.

SUMMARY:
This study investigates the implementation and effectiveness of the Family Check-Up 4 Health (FCU4Health) intervention in primary care settings for reducing cardiovascular disease risk in children. Through a hybrid type 3 cluster randomized factorial trial and innovative technology-based strategies integrated with Electronic Health Records, the study aims to enhance intervention fidelity and engagement. Results will inform scalable approaches to promote child and family health behaviors, improve parenting skills, and potentially reduce child BMI, contributing to significant public health impacts in addressing cardiovascular health disparities.

DETAILED DESCRIPTION:
The proposed implementation trial is a hybrid effectiveness-implementation type III design, with a primary focus on implementation strategies and outcomes. Eligible families include children aged 2-17 who are patients at Denova Integrated Healthcare. All families (n = 900-1200) will receive FCU4Health services from a Denova staff member trained in the intervention and supervised by FCU4Health experts. Following guidance from the ongoing Community Advisory Board, investigator's previous trials, and Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, implementation barriers were identified to scale-up and implementation strategies adopted for the trial: Lyssn fidelity support and Short Message Service (SMS) text messaging to promote program engagement.

Randomization to these strategies will occur at the care team level (n = 11-12) using a factorial design. Parent/caregivers and children at least 6 years of age will complete assessments at baseline, 6 months, 12 months, and 18 months.

Primary outcomes are fidelity and engagement (Aim 1a) and child health behaviors (Aim 1b). Investigators will also examine secondary outcomes including family health routines and parenting; conduct economic analyses (Aim 2); and examine the link between trajectories of improvement in health behaviors and improvements in BMI for subgroups related to baseline BMI, child developmental age group, race/ethnicity, language, and gender (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* BMI at or above 85 percentile for age and gender.

Exclusion Criteria:

* N/A

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Lyssn Fidelity Ratings | Up to 36 months
  Co-primary outcome of Aim 1: Fidelity to the motivational interviewing (MI) skills that are central to Family Check-Up 4 Health effects using the Lyssn automated coding platform. The system has been shown to be competitive with human coding using the Motivational Interviewing Skill Code (MISC) and the Motivational Interviewing Treatment Integrity Code (MITI 4). The Lyssn fidelity rating system consists of three dimensions: acceptance, empathy, and spirit, scored on a 7-point Likert scale. (1=low rating, 4=mid rating, 7=high rating). Lyssn scores are also convergent with human codings on the COACH observational rating system (see next measure).
Engagement in Family Check Up 4 Health (FCU4Health) (in-session caregiver engagement) | Up to 36 months
  Co-primary outcome of Aim 1: COACH rating system Parent In-Session Engagement Domain, 1-9 scale (1=low, 5=moderate, 9=high). Reliable and validly predictive of intervention outcomes.
Budget impact of implementation | Up to 48 months
  Co-Primary outcome of Aim 2: Cost capture survey based on time-driven activity-based costing methods and data from FCU4Health services provided.
Cost-effectiveness of FCU4Health | Up to 48 months
  Co-Primary outcome of Aim 2: Cost-effectiveness analysis using incremental cost-effectiveness ratios will be used to determine the value of each strategy as it relates to child BMI change and to implementation outcomes known to be related to intervention effects (e.g., fidelity). Data obtained via Cost capture survey based on time-driven activity-based costing methods and data from FCU4Health services provided.
Child Health Behaviors: Dietary Screener Questionnaire | Baseline, 6, 12, and 18 months
  Primary outcome of Aim 1b and Aim 3:
  National Health and Nutrition Examination Survey's Dietary Screener Questionnaire: 6 questions collect intake frequency of food (fruits, vegetables, fast food) and beverage choices (regular soda, 100 percent fruit juice, or sweetened fruit drinks, sports drinks, or energy drinks) during the past month. (i.e. During the past month, how often did you drink regular soda that contains sugar? Frequency of choices within past 2 weeks). The Dietary Screener Questionnaire has been shown to be a low burden food recall screener for specific dietary factors.
  This scale was administered in investigator's Centers for Disease Control and Prevention (CDC) funded trial and had good psychometrics as demonstrated using confirmatory factor analysis.
  Values range from 0-8. Never=0, 5-6 times per week=4, 6+per day=8. For food items, higher scores indicate healthier behaviors. For the beverage choices, lower scores indicate healthier behaviors.

SECONDARY OUTCOMES:
COACH Fidelity Rating System | Up to 36 months
  Conceptually accurate and adherent to the intervention model, Observant and responsive to the family's needs, Active in structuring the session, Careful when teaching and providing feedback, Helpful in building hope and motivation (COACH) observational rating system for FCU4Health consists of 5 domains, 1-9 scale (1=needs work, 5=competent work, 9=excellent work). Ratings have been found to be reliable and validly predict engagement and effectiveness outcomes.
Engagement (participation) in FCU4Health services | From enrollment to end of intervention at 18 months
  FCU4Health services received (attendance at intervention sessions, referrals completed)
Engagement in home practice | From enrollment to end of intervention at 18 month
  FCU4Health coordinator ratings of home practice using a rating scale found to be predictive of program outcomes, 1-9 scale. High Engagement (scores 7-9) Moderate Engagement (scores 4-6) Low Engagement (scores 1-3).
Engagement with the SMS text messaging platform | From enrollment to end of intervention at 18 month
  SMS Text messaging interactions (parent read/ response percentage rates)in the Configurable Assessment Messaging Platform for Interventions (CAMPI) platform *only for those in SMS study condition.
Child BMI - Percentage of the 95th percentile (BMIp95) | Baseline and 18 months
  Secondary outcome of Aim 1b and Aim 3: Children will be weighed using a portable electronic dual frequency bioelectrical impedance scale (Tanita SC-331SU). A portable stadiometer will take two height measurements, which are then averaged.
  A third measurement is taken if the ﬁrst two differ by more than one-eighth of an inch. Child BMI will be standardized by age and gender according to the CDC growth reference data for children, and percentage of the 95th percentile (BMIp95) will be calculated, as this is a more robust metric for assessing pediatric BMI change over time.
Reach of the intervention | Up to 36 months
  Secondary outcome of Aim 1: 1. Proportion of enrolled children/families (study participants) referred to FCU4Health / number eligible.
  2. Proportion of referred children/families engaged in the intervention / number eligible.
Normalisation MeAsure Development questionnaire | Month 6, Month 16, Month 24
  Secondary outcome of Aim 1: Acceptability, appropriateness, and feasibility of the implementation strategies.
  The Normalisation MeAsure Development questionnaire (NoMAD) comprises 23-items, concerned with: implementation (bringing a practice or practices into action); embedding (when a practice or practices may be routinely incorporated in everyday work); and integration (when a practice or practices are reproduced and sustained in the social matrices of an organization). A 5-point Likert scale is used for all responses (1=disagree, 3=neither agree nor disagree, 5=agree). Particularly relevant for evaluating implementation of technology in primary care.
Maintenance/Sustainability | Month 6, Month 16, Month 24
  Secondary outcome of Aim 1: Clinical Sustainability Assessment Tool: 21 items, 7 domains: Engaged Leadership and Staff; Engaged Stakeholders; Planning and Implementation; Workflow Integration; Monitoring and Evaluation; Organizational Context and Capacity; Outcomes and Effectiveness. A 7-point Likert scale is used for all domains (1=little or no extent, 4=some extent, 7=great extent). Reliable and valid.
Parenting Skills: Incentives and Encouragement | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Positive Behavior Support: Incentives and Encouragement survey consists of 4 items and uses a 5-point Likert scale (0=never, 3=sometimes, 4=very often). Higher scores indicating better positive behavior supports in the domain of parent incentives and encouragement.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Proactive Parenting | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Positive Behavior Support: Proactive Parenting survey consists of 7 items and uses a 5-point Likert scale (0=never, 3=sometimes, 4=very often). Higher scores indicating better positive behavior supports in the domain of proactive parenting.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Parenting Warmth | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Relationship Quality: Parenting Warmth survey consists of 5 items and uses a 5-point Likert scale (1=not at all, 3=somewhat true, 4=very true). Higher scores indicating better ratings of relationship quality in the domain of parenting warmth.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Parent-Child Conflict | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Relationship Quality: Parent-Child Conflict survey consists of 10 items and uses a 5-point Likert scale (1=not at all, 3=somewhat true 4=very true). Lower scores indicating better ratings of relationship quality in the domain of parent-child conflict.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Quality Time | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Relationship Quality: Quality Time survey consists of 6 items and uses a 5-point Likert scale (0=never, 3=sometimes, 4=very often). Higher scores indicating better ratings of relationship quality in the domain of parent-child quality time.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Monitoring and Limit Setting | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Monitoring and Limit Setting survey consists of 7 items and uses a 5-point Likert scale (0=never, 3=sometimes, 4=very often). Higher scores indicating better parent monitoring and limit setting.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Parenting Skills: Negative Parenting Behaviors | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b:
  The Negative Parent Behaviors survey consists of 5 items and uses a 5-point Likert scale (0=never, 3=sometimes, 4=very often). Lower scores indicating better ratings of parent behaviors.
  This domain has minor age- appropriate variations for ages 2-5 years, 6-12 years, and 13+ years that are valid and reliable.
Family Health Routines: Mealtime | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b: Mealtime Parenting Scale: 5 items using a 5-point Likert scale (0=almost never, 2=sometimes, 4=nearly always). Scale was administered in investigator's CDC-funded trial and had good psychometrics as demonstrated using confirmatory factor analysis.
Family Health Routines: Media | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b: Media Parenting Scale: 3 items using a 5-point Likert scale (0=almost never, 2=sometimes, 4=nearly always). Scale was administered in investigator's CDC-funded trial and had good psychometrics as demonstrated using confirmatory factor analysis.
Family Health Routines: Sleep | Baseline, 6, 12, and 18 months
  Secondary outcome of Aim 1b: Sleep Parenting Scale 8 items from existing scales that have shown high validity and reliability (i.e., Children's Sleep Wake Scale, Children's Sleep Hygiene Scale, Parental Interactive Behaviour Scale, Brief Infant Sleep Questionnaire and the Sleep Environment Scale). Uses a 5-point Likert scale (0=almost never, 2=sometimes, 4=nearly always). Scale was administered in investigator's CDC-funded trial and had good psychometrics as demonstrated using confirmatory factor analysis.

OTHER OUTCOMES:
Satisfaction with FCU4Health Parent Service | Month 12 and Month 18 surveys to parents
  FCU4Health Parent Service Satisfaction Survey. 8 items (α>.95). Adapted from the validated Client Satisfaction Questionnaire. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Satisfaction with FCU4Health Parent-Coordinator | Month 12 and Month 18 surveys to parents
  Parent-Coordinator Collaboration, Systemic Awareness, and Negative Feelings subscales of the Parent Experience of Assessment Survey (12 items total; α>.75) The survey uses a 5-point Likert scale (1=Strongly Disagree, 3=Neutral, 5=Strongly Agree) with the higher number indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Cady Berkel, Ph.D., Principal Investigator — Arizona State University; Justin D Smith, Ph.D., Principal Investigator — University of Utah
Locations (1):
- Denova Integrated Healthcare, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No